CLINICAL TRIAL: NCT04123093
Title: Safety and Efficacy of the Noxsano Wound Care Bandage: A First in Human Study
Brief Title: Safety and Efficacy of the Noxsano Wound Care Bandage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to rigorous inclusion criteria and the constraints brought on the health care system from the COVID 19 pandemic which adversely effected enrollment, the sponsor and collaborator have decided to halt enrollment and officially close out the study.
Sponsor: OhioHealth (Other)
Collaborators: Noxsano, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1331496
Record Dates: First submitted 2019-09-18; First posted 2019-10-10 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Wound Heal; Peripheral Artery Disease; Ulcer, Leg; Ulcer Foot; Diabetic Foot Ulcer; Arterial Insufficiency
MeSH Terms: conditions — Peripheral Arterial Disease; Leg Ulcer; Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The study has two interventions: (1) Noxsano Bandage (Healthy Volunteers) and (2) Noxsano Bandage (Wound Care). Each intervention is associated with a separate group of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): The initial phase of the study is designed to determine the safety of the study device, the Noxsano Bandage, in healthy volunteers without wounds.
  Interventions: Device: Noxsano Bandage (Healthy Volunteers)
- Wound care (Experimental): The second phase of the study is designed to determine the effectiveness of the study device in wound healing in subjects with active wounds.
  Interventions: Device: Noxsano Bandage (Wound Care)

INTERVENTIONS:
Device: Noxsano Bandage (Healthy Volunteers) — Healthy volunteers will wear the study device (Noxsano Bandage) for 3 consecutive days (up to 72 hours), followed by weekly visits for 4 weeks of observation for tolerance, side effects, and/or adverse reactions.
  Arms: Healthy Volunteers
Device: Noxsano Bandage (Wound Care) — Wound care subjects will have weekly study device (Noxsano Bandage) applications to a specific ulceration. For subjects that exhibit any reduction in wound surface area, this application will occur until the wound is healed, or for up to 3 months (whichever occurs first). For subjects that do not exhibit any reduction in wound size at 2 months, application will stop and standard treatment protocols will be pursued. At the conclusion of the treatment window (up to 3 months), subjects will be followed every 3 months for 12 consecutive months for observation of late side effects or adverse reactions (3 months of active treatment, 12 months of follow-up observation, 15 months total).
  Arms: Wound care

SUMMARY:
This study is a prospective, interventional, non-randomized study designed to assess the safety and efficacy of the Noxsano Bandage (study device) in healthy subjects and wound care subjects with a diabetic lower extremity ulceration and/or arterial insufficiency lower extremity ulceration.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Subjects must meet all of the following criteria to be eligible for enrollment:

1. Subject is ≥ 18 and < 80 years of age.
2. Subject is white, black or African American
3. Subject has provided written informed consent.
4. Subject is willing to comply with study follow-up requirements.
5. Subject has intact skin on lower extremities.

Group 2: Subjects must meet all of the following criteria to be eligible for enrollment:

1. Subject is ≥ 18 and < 80 years of age.
2. Subject has a baseline wound surface area of < 25 cm2.
3. Subject has provided written informed consent.
4. Subject is willing to comply with study follow-up requirements.
5. Subject with at least one of the following:

   1. Diabetic lower extremity ulceration with a hemoglobin A1c (HgbA1c) value ≤ 9.0, drawn within 3 months prior to study participation , and/or
   2. Arterial insufficiency lower extremity ulceration with a post-revascularization ankle-brachial index (ABI) value of ≥ 0.40 and ≤ 0.80 on the involved extremity, performed within 3 months prior to study participation1, and/or
   3. Diabetic and/or arterial insufficiency lower extremity ulceration deemed in-eligible for revascularization with 3 months prior to study participation

Exclusion Criteria:

Group 1: Subjects will be excluded from the trial if any of the following criteria are met:

1. Subject is < 18 or ≥ 80 years of age.
2. Subject has a history of diabetes, arterial insufficiency, or osteomyelitis.
3. Subject has a known hypersensitivity to adhesives.
4. Subject is on any prescription medications, including contraceptives. Due to the short duration of the procedure period (3 days), subjects who initiate prescription medications during study participation will continue in the study.
5. Subject is pregnant, plans to become pregnant during the study period, or is breastfeeding.
6. Subject is non-English speaking or reading.
7. Subject is unable to give informed consent. -

Group 2: Subjects will be excluded from the trial if any of the following criteria are met:

1. Subject is < 18 or ≥ 80 years of age.
2. Subject has a baseline wound surface area of ≥ 25 cm2.
3. Subject has a plantar wound.
4. Subject with diabetes with an HgbA1c value of > 9.0, drawn within 3 months prior to study participation . Subject with arterial insufficiency with an ABI value of < 0.40 or > 0.80, performed within 3 months prior to study participation .
5. Subject with osteomyelitis contiguous with the ulceration treatment site.
6. Subject with peripherally-inserted central catheter (PICC) line antibiotic treatment within the previous 6 months.
7. Subject requiring any type of amputation on the treatment limb within 3 months prior to study participation.
8. Subject with a known hypersensitivity to adhesives.
9. Subject is on active steroid therapy (does not include inhaled steroids).
10. Subject is pregnant, plans to become pregnant during the study period, or is breastfeeding.
11. Subject is non-English speaking or reading.
12. Subject is unable to give informed consent.
13. Subject is currently enrolled in another interventional study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Silver, DO, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is designed to enroll into each arm sequentially. Therefore healthy subjects are enrolled first and once they have completed follow-up, wound care patients are eligible for enrollment.
Groups:
- Healthy Volunteers: Healthy volunteers with no skin wounds and who are not taking any prescription medications.
- Wound Care: Subjects with a lower extremity ulceration attributed to diabetes and/or arterial insufficiency.
Period: Phase 1
Arm/Group | Healthy Volunteers | Wound Care
Started | 11 | 0
Baseline Visit | 10 | 0
Completed | 10 | 0
Not Completed | 1 | 0
Not completed — Subject did not show up for baseline visit and was replaced | 1 | 0
Period: Phase 2
Arm/Group | Healthy Volunteers | Wound Care
Started | 0 | 2
Baseline Visit | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Wound Care | Total
Number analyzed (Participants) | 10 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants] — Age at baseline visit
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 0 | 9
    >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (13.4) | 69.5 (0.5) | 44.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 2 | 12
Body Mass Index [Mean (Standard Deviation); unit: kilograms pre meter squared] — Data collected at the initial study visit, prior to Noxsano bandage application Population: Body Mass Index (BMI) data was not collected for healthy volunteers
  kilograms pre meter squared
    number analyzed (Participants) | 0 | 2 | 2
    (all) |  | 29.8 (1.0) | 29.8 (1.0)
Height [Mean (Standard Deviation); unit: centimeters] — Data collected at the initial study visit, prior to Noxsano bandage application Population: Height data was not collected for healthy volunteers
  centimeters
    number analyzed (Participants) | 0 | 2 | 2
    (all) |  | 175.3 (5.1) | 175.3 (5.1)
Hemoglobin A1c [Mean (Standard Deviation); unit: mmol/mol] — Most recent hemoglobin A1C reading Population: Hemoglobin A1c measurements were not collected for health volunteers
  mmol/mol
    number analyzed (Participants) | 0 | 2 | 2
    (all) |  | 7.8 (0.7) | 7.8 (0.7)
Medical History [Number; unit: participants] — Number of participants diagnosed with diabetes, vascular disease hypertension, and end stage renal disease
  participants
    Diabetes | 0 | 2 | 2
    Vascular Disease | 0 | 2 | 2
    End Stage Renal Disease | 0 | 2 | 2
Concomitant Medications [Number; unit: participants] — List of medications collected at the initial study visit, prior to Noxsano bandage application
  participants
    atorvastatin | 0 | 2 | 2
    amlodipine | 0 | 1 | 1
    clopidogrel | 0 | 1 | 1
    hydrocodone -acetaminophen | 0 | 1 | 1
    hydrochlorothiazide | 0 | 1 | 1
    gabapentin | 0 | 1 | 1
    lidocaine cream | 0 | 1 | 1
    lisinopril | 0 | 1 | 1
    losartan | 0 | 1 | 1
    metformin | 0 | 2 | 2
    metoprolol | 0 | 1 | 1
    rivaroxaban | 0 | 1 | 1
    valsartan-hydrochlorothiazide | 0 | 1 | 1
    potassium chloride SA | 0 | 1 | 1
    spironolactone | 0 | 1 | 1
    Vitamin C | 0 | 1 | 1
    Vitamin D3 | 0 | 1 | 1
Smoking History [Number; unit: participants] — History of tobacco product use. Population: Smoking history data was not collected for healthy volunteers.
  participants
    Current Smoker: number analyzed (Participants) | 0 | 2 | 2
    Current Smoker |  | 0 | 0
    Former Smoker: number analyzed (Participants) | 0 | 2 | 2
    Former Smoker |  | 1 | 1
    Never Smoked: number analyzed (Participants) | 0 | 2 | 2
    Never Smoked |  | 1 | 1
Weight [Mean (Standard Deviation); unit: kilograms] — Weight collected at the initial study visit, prior to the Noxsano bandage application. Population: Weight was not collected for healthy volunteers
  kilograms
    number analyzed (Participants) | 0 | 2 | 2
    (all) |  | 82.1 (1.8) | 82.1 (1.8)
Wound Care [Number; unit: participants] — Standard wound care techniques that were performed on the patient prior to study initiation Population: This measurement does not apply to healthy volunteers as they do not have skin wounds.
  participants
    Debridement: number analyzed (Participants) | 0 | 2 | 2
    Debridement |  | 2 | 2
    Dermagraft: number analyzed (Participants) | 0 | 2 | 2
    Dermagraft |  | 1 | 1
Wound Size [Median (Full Range); unit: centimeters squared] — Wound area calculated by length times width Population: Wound size does not apply to healthy volunteers as they do not have wounds.
  centimeters squared
    number analyzed (Participants) | 0 | 2 | 2
    (all) |  | 8.98 [2.2 to 15.75] | 8.98 [2.2 to 15.75]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events - Healthy Volunteers
Description: Adverse events related to the Noxsano bandage will be assessed using a safety and adverse reactions questionnaire that includes questions for the subject regarding tolerance, side effects, and adverse events.
Time Frame: 4 weeks post-bandage removal
Population: Number of participants with an adverse event four weeks post bandage removal
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 10
Participants | 3

2. Primary Outcome: Wound Surface Area
Description: Wound surface area will be measured using a horizontal and vertical measurement taken in centimeters (cm) using a standard ruler. These measurements are used to calculate wound area in centimeters squared (cm2).
Time Frame: change in baseline wound area at 2 months
Population: The study was not completed and data for this outcome were not collected
Arm/Group | Wound Care
Number analyzed (Participants) | 0

3. Secondary Outcome: Adverse Events - Wound Care Subjects
Description: as for outcome 1
Time Frame: 12 months post-treatment
Population: The study was not completed and these data were not collected
Arm/Group | Wound Care
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 4 weeks for Healthy Volunteers and up to 13 months for Wound Care participants.
Description: A questionnaire about adverse events was administered to each patient. The questionnaire asked about adverse reactions related to the skin and application site, systemic reactions, infections, and allergic reactions.
Arm/Group | Healthy Volunteers | Wound Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/2
Other Adverse Events (participants affected / at risk) | 7/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=10) | Wound Care (N=2)
Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Volunteers (N=10) | Wound Care (N=2)
itchy skin (Skin and subcutaneous tissue disorders) | 7 | 1
dry dkin (Skin and subcutaneous tissue disorders) | 5 | 1
pain (Skin and subcutaneous tissue disorders) | 2 | 1
red skin (Skin and subcutaneous tissue disorders) | 1 | 1
swollen skin (Skin and subcutaneous tissue disorders) | 2 | 1
bruise (Skin and subcutaneous tissue disorders) | 2 | 0
skin discoloration (Skin and subcutaneous tissue disorders) | 5 | 0
skin flaking (Skin and subcutaneous tissue disorders) | 1 | 0
skin darkening (Skin and subcutaneous tissue disorders) | 0 | 1
pressure sores (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04123093/Prot_SAP_000.pdf
  • Informed Consent Form: Healthy Volunteer Consent (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04123093/ICF_001.pdf
  • Informed Consent Form: Wound Care Patient Consent (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04123093/ICF_002.pdf